CLINICAL TRIAL: NCT05626673
Title: Feasibility and Preliminary Efficacy of Using a Faith and Prayer Mobile App, Pray.Com, on Mental Health and Well-being in a Sample of Racial/Ethnic Minorities
Brief Title: Exploring the Experience of Using a Prayer Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biola University (Other)
Responsible Party: Principal Investigator, Todd Hall, Professor, Biola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: F22-013
Record Dates: First submitted 2022-11-08; First posted 2022-11-25 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: No Specific Condition. Feasibility of Mobile App

STUDY DESIGN:
Intervention Model Description: Participants will be provided access to the Pray.com app and directed to use it for at least 5 minutes per day for at least 5 times per week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prayer app (Experimental): Participants will be given the Pray.com app and directed to use it daily.
  Interventions: Behavioral: Prayer app

INTERVENTIONS:
Behavioral: Prayer app — Participants will be given the Pray.com app and directed to use it daily.

SUMMARY:
The goal of this clinical trial is to explore the feasibility and preliminary effects of using Pray.com on spiritual well-being and mental health symptoms in racial/ethnic minority adults. The main question it aims to answer is: What are the feasibility and preliminary effects of using Pray.com on spiritual well-being and mental health (stress, depressive and anxiety symptoms) in racial ethnic minority adults (i.e., individuals who identify as Black/African American, Latinx/Hispanic, Asian/Pacific Islander, Native American, or Multiracial)?

Participants will be given the Pray.com app and directed to use it daily. Participants will complete measures at baseline (i.e., time 1) and four-weeks (i.e., time 2). A smaller subset of participants will be asked to participate in a qualitative interview.

DETAILED DESCRIPTION:
Participants (N = 75) will be recruited through social media and various Christian organizations that serve racial/ethnic minorities. Participants will be over the age of 18 and identify as a racial/ethnic minority (i.e., individuals who identify as Black/African American, Latinx/Hispanic, Asian/Pacific Islander, Native American, or Multiracial). Participants also must be willing to participate in a study that involves engaging in a regular Christian religious practice and are willing to download the Pray.com app.

Eligible participants will be given the Pray.com app and directed to use it daily. Participants will complete measures at baseline (i.e., time 1) and four-weeks (i.e., time 2). At the end of the study participants will be randomly asked to participate in an interview (N = 15) which will take no longer than 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Identify as a racial/ethnic minority (e.g., Black/African American, Latinx/Hispanic, Asian/Pacific Islander, Native American, Multiracial).
* Own a smart phone and be willing to download a mobile app.
* Willing to engage in a Christian-based religious practice on a mobile app.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hall, PhD, Principal Investigator — Biola University
Locations (1):
- Biola University, La Mirada, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants were provided access to the Pray.com app at no cost and directed to use 5 minutes per day for at least 5 days per week.
Period: Overall Study
Arm/Group | Intervention
Started | 77
Completed | 72
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Prayer App
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Black or African American | 65
  Race and Ethnicity: American Indian/Native American | 6
  Race and Ethnicity: Alaskan Native | 0
  Race and Ethnicity: Asian or Asian American | 1
  Race and Ethnicity: Native Hawaiian or Pacific Islander | 2
  Race and Ethnicity: Latina/Latino/Hispanic | 3
Perceived Stress Scale-10 [Mean (Standard Deviation); unit: units on a scale] | 2.72 (.66)
Hospital Anxiety and Depression Scale-Anxiety [Mean (Standard Deviation); unit: units on a scale] | 1.12 (.59)
Hospital Anxiety and Depression Scale-Depression [Mean (Standard Deviation); unit: units on a scale] | .84 (.53)
Religious Commitment Inventory-10 [Mean (Standard Deviation); unit: units on a scale] | 3.84 (.71)
Spiritual Well-Being Scale [Mean (Standard Deviation); unit: units on a scale] | 4.47 (.80)
Satisfaction with Life Scale [Mean (Standard Deviation); unit: units on a scale] | 4.68 (1.26)
Multiethnic Identity Measure [Mean (Standard Deviation); unit: units on a scale] | 3.96 (.63)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Mobile App
Description: 9 questions created for the present study, Minimum value: 1, Maximum value: 5, Higher scores reflect higher acceptability (i.e., better outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prayer App: Participants were provided access to the Pray.com app at no cost and directed to use for it at least 5 minutes per day for at least 5 days per week.
  Prayer app: Participants were provided access to the Pray.com app at no cost and directed to use for it at least 5 minutes per day for at least 5 days per week.
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale
  Satisfaction | 4.5 (.69)
  Intent to continue use | 4.47 (.71)
  Relevance in improving mental health | 4.14 (.74)
  Relevance in improving spiritual life | 4.42 (.88)
  Racial/ethnic identity well-represented | 4.29 (.74)
  Content good fit with racial/ethnic identity | 4.15 (.85)
  Content good fit with cultural worldview | 4.29 (.76)
  App good fit with religious beliefs or worldview | 4.25 (.87)
  App good fit with cultural identity or worldview | 4.11 (.87)

2. Primary Outcome: Demand for Mobile App
Description: 3 questions created for the present study, Minimum value: 1, Maximum value: 5, Higher scores reflect higher demand (i.e., better outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prayer App: Participants were provided access the Pray.com app at no cost and directed to use it for at least 5 minutes per day for at least 5 days per week.
  Prayer app: Participants were provided access the Pray.com app at no cost and directed to use it for at least 5 minutes per day for at least 5 days per week.
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale
  Frequency of use | 3.11 (.74)
  Interest in future use | 4.31 (.73)
  Perceived demand within participants' religious community | 4.29 (.83)
  Perceived demand within participants' cultural community | 4.11 (.82)

3. Primary Outcome: Practicality of Mobile App
Description: 5 questions created for the present study, Minimum value: 1, Maximum value: 5, Higher scores reflect higher practicality (i.e., better outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prayer App: Participants were provided access to the Pray.com app and directed to us it for at least 5 minutes per day for at least 5 days per week.
  Prayer app: Participants were provided access to the Pray.com app and directed to us it for at least 5 minutes per day for at least 5 days per week.
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale
  Difficulty of use | 1.76 (.90)
  Ability to use and navigate app | 4.35 (.70)
  Perceived cost of the app | 2.46 (.86)
  Ease of paying monthly fee | 2.35 (.97)
  Willingness to pay monthly fee | 4.14 (.83)

4. Primary Outcome: Minutes of App Use
Description: How many minutes did the participant use the mobile app?
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Prayer App: Participants were provided access to the Pray.com app and directed to use it for at least 5 minutes per day for at least 5 times per week.
  Prayer app: Participants were provided access to the Pray.com app and directed to use it for at least 5 minutes per day for at least 5 times per week.
Arm/Group | Prayer App
Number analyzed (Participants) | 72
minutes | 45.83 (111.90)

5. Secondary Outcome: Spiritual Well-being Scale
Description: Minimum value: 1, Maximum value: 6, Higher scores reflect higher spiritual well-being (i.e., better outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale | 4.89 (.83)

6. Secondary Outcome: Satisfaction With Life Scale
Description: Minimum value: 1, Maximum value: 6, Higher scores reflect higher satisfaction with life (i.e., better outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale | 5.31 (.97)

7. Secondary Outcome: Religious Commitment Inventory
Description: Minimum value: 1, Maximum value: 5, Higher scores reflect higher religious commitment (i.e., better outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale | 4.01 (.61)

8. Secondary Outcome: Multiethnic Identity Measure
Description: Minimum value: 1, Maximum value: 5, Higher scores reflect higher ethnic identity (i.e., better outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale | 4.09 (.58)

9. Secondary Outcome: Perceived Stress Scale
Description: Minimum value: 0, Maximum value: 5, Higher scores reflect higher stress (i.e., worse outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale | 2.52 (.71)

10. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: Minimum value: 0, Maximum value: 3, Higher scores reflect higher anxiety/depression (i.e., worse outcome)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prayer App
Number analyzed (Participants) | 72
units on a scale
  Anxiety | .98 (.58)
  Depression | .70 (.57)

11. Primary Outcome: Days of App Usage
Description: How many days did the participant use the mobile app?
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Prayer App
Number analyzed (Participants) | 72
Days | 5.77 (8.19)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Prayer App
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-11-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05626673/Prot_SAP_ICF_000.pdf